CLINICAL TRIAL: NCT04508959
Title: A Rapid Research Platform to Inform Prevention & Improve the Clinical Management of COVID-19 Illness for Priority Older Adult Groups: The McMaster Multi-regional Hospital Coronavirus Registry
Brief Title: The McMaster Multi-Regional COVID-19 Hospital Case Registry
Acronym: COREG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Hamilton Academic Health Sciences Organization (Other); Grand River Hospital (Other); Niagara Health System (Other); St. Mary's General Hospital (Unknown); Hamilton Health Sciences Corporation (Other); St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Andrew Costa, Associate Professor and Schlegel Chair in Clinical Epidemiology & Aging, McMaster University
Other Study IDs: 172754
Record Dates: First submitted 2020-08-10; First posted 2020-08-11 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Coronavirus Infection; Coronavirus; SARS-CoV-2 Infection; Covid19
Keywords: Registry
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Screened patients: All individuals screened using the hospital's microbiology laboratory.
- Outpatient (Emergency Department) cases: All individuals seen in the emergency department who test positive for COVID-19.
- Inpatient (General Medical or Intensive Care) cases: All individuals admitted to a general or intensive care bed who test positive for COVID-19.

SUMMARY:
The McMaster Multi-Regional Hospital Coronavirus Registry (COREG) is a platform that is collecting detailed case data on laboratory confirmed COVID-19 hospital inpatients and outpatients. The COREG platform will provide rapid high-quality evidence to improve the prevention and clinical management of COVID-19 for older adults in Canada, and internationally. The COREG platform will also provide researchers and partners with complete regional level clinical data on COVID-19 cases to inform rapid decision-making and projections, sub-studies, extensions, and linkage for all affected populations.

DETAILED DESCRIPTION:
Rationale: The novel coronavirus disease of 2019 (COVID-19) is a rapidly evolving pandemic, which poses a major and ongoing threat to health and the health system both globally and locally. While there have been country-specific case series that have offered some guidance on interventions that may be effective; applying them to local settings is problematic, given differences in population density, demographics (including vulnerable sub-populations), economic and political capacity. To this end, local data is needed to better inform on the timing and implementation of specific and targeted interventions to mitigate the spread and impact of the virus immediately, and thereafter. Near real-time information can greatly inform efforts and decisions needed to address resource allocation in response to the dynamic pandemic.

Objectives: The Investigators' aim is to collect data on the impact and burden of COVID-19 that can inform and support real-time local clinical and policy decisions. Specifically, the objectives are to: 1) Create a COVID-19 admission case registry as a local research and quality improvement platform for the COVID-19 pandemic; and 2) Collect data that can inform local pandemic decisions and evaluation, including incidence, vulnerability, complications, and clinical course of COVID-19 patients.

Methods: The investigators have established the McMaster Coronavirus (COVID-19) Registry (COREG), an ISARIC-WHO compatible, comprehensive platform that facilitates uniform data collection of COVID-19. COREG is an extension of the ISARIC-WHO case report form (CRF) designed to capture local information on transmission, disease- burden, course, and outcomes of COVID-19 cases from all COVID-19 charting hospitals in the Waterloo, Hamilton, and Niagara Regions of Ontario, Canada (Population > 1,500,000). COREG is a comprehensive patient registry based retrospective data collection on all suspected and confirmed COVID-19 cases (according to the ISARIC definition) admitted to St. Joseph's Healthcare Hamilton (SJHH), Hamilton Health Sciences (HHS), Grand River Hospital, St. Mary's General Hospital, and the Niagara Health System. The registry includes data abstracted from existing chart data generated during routine clinical care. A waiver of informed consent is granted. Data categories to be collected follow the ISARIC-WHO CRF (https://isaric.tghn.org/covid-19-clinical-research-resources/) and include demographics, co-morbidities, pre-admission medications, signs and symptoms, diagnostic results, in-hospital interventions and health outcomes (medical complications during hospitalization including ICU and death). Cases are identified by the Infection Prevention and Control (IPAC) at each site and records will be accessed remotely and securely by research and medical staff. Extracted data are stored in a secure McMaster hosted REDCap and data server. Data collectors undergo a standardized training. Weekly governance meetings occur between the data collectors, operational leads and clinical site lead at each site to discuss, address and resolve any barriers and inconsistences in data collection and advance the scientific agenda.

Impact: COREG ensures that COVID-19 data collected are standardized and robust and will have a meaningful impact on local decision-making, while also being comparable internationally. COREG will shape consensus recommendations on inpatient management of hospitalized patients with COVID-19. It will be invaluable to local and global research efforts, since linkage to tissue biobanks and other administrative databases can be easily performed to address questions on pathophysiology, long-term outcomes and healthcare burden.

ELIGIBILITY:
Inclusion Criteria:

* Persons tested positive for SARS-CoV-2 using hospital facilities
* Patients seen or admitted with confirmed COVID-19 to the hospital

Exclusion Criteria:

* The pragmatic nature of the registry warrants the broadest inclusion criteria that are feasible. In keeping with the pragmatic nature of this registry, no exclusions are introduced.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Persons tested positive for SARS-CoV-2 using hospital facilities
  * Patients seen or admitted with confirmed COVID-19 to the hospital
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-04-15 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Serious COVID-19 infection | through study completion, an average of 1 year
  Defined as symptomatic hospital outpatients with laboratory confirmed SARS-CoV-2 (based on the ISARIC definition) through the COREG platform.
Severe infection (requiring admission) | through study completion, an average of 1 year
  Defined as persons admitted with laboratory confirmed SARS-CoV-2 (based on the ISARIC definition) available through the COREG platform. We will also conduct sub analyses of hospital acquired COVID-19 also captured in the COREG platform.
COVID-19 related death | through study completion, an average of 1 year
  Defined as persons who died with laboratory confirmed SARS-CoV-2 (based on the ISARIC definition) available through the COREG platform.

SECONDARY OUTCOMES:
Length of stay | through study completion, an average of 1 year
  Days from admission to discharge.
Complications | through study completion, an average of 1 year
  New or increased severity of conditions and syndromes from pre-morbid state.
Intensive interventions | through study completion, an average of 1 year
  Rate of intensive interventions during hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca J Kruisselbrink, MD, MPH, FRCPC, Principal Investigator — McMaster University; MyLinh Duong, MBBS, MSc, FRACP, Principal Investigator — McMaster University; Terence Ho, MD, FRCP, Principal Investigator — McMaster University; Andrew P Costa, PhD, Principal Investigator — McMaster University; Marla Beauchamp, PhD, Principal Investigator — McMaster University; Jennifer Tsang, MD, PhD, FRCPC, Principal Investigator — McMaster University
Locations (5):
- Canada (5):
  - Hamilton General Hospital, Hamilton, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Grand River Hospital, Kitchener, Ontario
  - St. Mary's General Hospital, Kitchener, Ontario
  - Niagara Health System, St. Catharines, Ontario

IPD SHARING:
Plan to Share IPD: Yes
WHO-ISARIC COVID-19 database (https://isaric.tghn.org/covid-19-clinical-research-resources/).
Time Frame: Entire registry